CLINICAL TRIAL: NCT03045718
Title: Effects of Horticultural Therapy on Elderly at Risk of Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Parks Board, Singapore (Other); Ministry of Health, Singapore (Other Government); Ministry of National Development, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016/00949
Record Dates: First submitted 2017-02-05; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Horticultural Therapy; Dementia
Keywords: Horticultural Therapy; Dementia; Randomized Controlled Trial; Elderly; Prevention
MeSH Terms: conditions — Dementia | interventions — Horticultural Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horticultural Therapy (Experimental): Horticultural Therapy will consists of 1 hour sessions, weekly for 9 months, to engage subjects in gardening-based activities.
  Interventions: Behavioral: Horticultural Therapy
- Waitlist Control (Other): The control group will be placed on a waiting list and only be contacted for assessments. They will receive the same Horticultural Therapy intervention after the active treatment group at a later date.
  Interventions: Behavioral: Horticultural Therapy

INTERVENTIONS:
Behavioral: Horticultural Therapy — The Horticultural Therapy intervention will be delivered by trained facilitators at the Therapeutic Garden at Hort Park, and consists of 1 hour sessions weekly for 9 months. The Horticultural Therapy program is designed to stimulate the senses through interaction with the tasks and the environment, promote social interaction and also to promote a sense of self-worth through completion of projects. It encompasses a range of activities including general gardening and also project-based craft activities.

SUMMARY:
The objective of this study is to determine whether horticultural therapy would improve the psychological well-being older adults who are at risk of memory (cognitive) decline. 100 elderly subjects who are at risk of cognitive decline will be randomized into the active horticultural therapy or to the waitlist control group. Sessions will be conducted weekly for 9 months, and participants will be assessed at 3 time-points: at the start of the study, at 3 months and at 9 months.

It is hypothesized that participants who undergo horticultural therapy will perform better on neuropsychological tests when compared to control, and that they will have improved psychological well-being and functional outcomes.

DETAILED DESCRIPTION:
Study participants comprise of community-dwelling elderly who are at risk of developing dementia, and will be selected from consenting participants from an existing community cognitive screening program.

This is an intervention study where 100 subjects will be randomized into an active horticultural therapy group, or a waitlist control group. Baseline demographic data will be collected at the start of the study. Assessments will be done at the start, at 3 months and at 6 months, which will include neuropsychological tests of cognitive functioning, psychological tests for depression and anxiety, assessment of psychosocial well-being, and tests of functional status.

The Horticultural Therapy intervention will be delivered by trained facilitators at the Therapeutic Garden at Hort Park, and consists of 1 hour sessions weekly for 9 months. The Horticultural Therapy program is designed to stimulate the senses through interaction with the tasks and the environment, promote social interaction and also to promote a sense of self-worth through completion of projects. It encompasses a range of activities including general gardening and also project-based craft activities.

The control group will be placed on a waiting list and only be contacted for assessments. They will receive intervention after the active treatment group at a later date.

ELIGIBILITY:
Inclusion Criteria:

1. Community-living elderly aged 60 years and above, AND 2.

1. Mild Cognitive Impairment based on clinical history and neuropsychological test scores (Z score <0 and >-1.5), OR
2. Subjective Memory Impairment based on self-report, OR (C) 2 or more risk factors for dementia such as family history, cerebrovascular disease, and cardiovascular risk factors

Exclusion Criteria:

1. Existing diagnosis of dementia, OR
2. Comorbid major mental illness (such as Major Depressive Disorder and Psychosis), OR
3. Severe or unstable life-limiting medical illness, OR
4. Severe physical impairment precluding participation in Horticultural Therapy

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Clinical Dementia Rating (CDR) at baseline and at 9 months | Baseline, 9 months
  Clinical Dementia Rating (CDR ) is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care.
Changes in Colour Trails Tests (CTT) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  Colour Trails Tests (CTT) 1 and 2 assesses sustained attention and sequencing.
Changes in Digit Span Task scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  Digit Span Task, which consists of a Digit Span Forward (DSF) and a Digit Span Backward (DSB) task is used to assess attention and verbal working memory.
Changes in Rey Auditory Verbal Learning Test (RAVLT) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  Rey Auditory Verbal Learning Test (RAVLT) evaluates declarative verbal learning and memory.
Changes in Block Design scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  Block Design is a subtest that is administered as part of several of the Wechsler Intelligence tests, and it primarily measures visual-spatial and organizational processing abilities, as well as non-verbal problem-solving skills
Changes in Semantic Verbal Fluency scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  Semantic Verbal Fluency assess lexical knowledge and semantic memory organization.

SECONDARY OUTCOMES:
Changes in Zung Self-Rating Depression Scale (SDS) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  The SDS (Zung, 1965) is a 20-item quantitative measurement of symptoms of depression. Participants rate each item regarding how they felt during the week preceding using a 4-point scale that ranges from 1 (a little of the time) to 4 (most of the time). A total raw score computed by summing the scores on the individual items will be converted into a percentage (the SDS index); the higher the SDS index, the greater the severity of depressive symptoms. Several studies have established the SDS as a reliable and valid instrument for measuring depressive symptoms (Biggs et al., 1978; Gabrys and Peters, 1985; Agrell and Dehlin, 1989).
Changes in Zung Self-Rating Anxiety Scale (SAS) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  The SAS (Zung, 1971) will be used to measure anxiety of the participants in the preceding week. It is a 20-item self-report assessment designed to measure anxiety levels, based on cognitive, autonomic, motor and central nervous system symptoms. Each question is scored on a Likert-type scale of 1-4 (a little of the time) to (most of the time). Some questions are negatively worded to avoid the problem of set response. Overall assessment is done by total score. The total raw scores range from 20-80. The raw score then needs to be converted to an "Anxiety Index" score; the higher the SAS index, the greater the severity of depressive symptoms.
Changes in Ryff's Scales of Psychological Well-being scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  The Ryff Scales of Psychological Well-Being (Ryff and Singer, 1998) is an 18-item questionnaire which reflects the six areas of psychological well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Respondents rate statements on a scale of 1 to 6, with 1 indicating strong disagreement and 6 indicating strong agreement.
Changes in Friendship Scale (FS) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  Social connectedness scale will be measured using the Friendship Scale (Hawthorne, 2006). It is a 6-item questionnaire that measures both social isolation and social connectedness. Participants were asked to rate the frequency in which each statement describes them during the past four weeks on a 5-point Likert scale ranging from 0 (almost always) to 5 (not at all). Total scores were computed by summing the scores on the individual items and ranged from 0 to 24, with higher scores indicating higher level of social connectedness. The Friendship Scale was developed as a short, user-friendly, stand alone scale measuring perceived social isolation. It was validated with older adults with excellent internal structures, reliability and validity (Hawthorne, 2006; Hawthorne, 2008).
Changes in EuroQol Five Dimensions Questionaire (ED-5D-3L) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  The E5-5D-3L is a standardized instrument for measuring general health status, which consists of 5 questions and a visual analog scale - which is a self-rating scale ranging from zero (0) to one hundred (100) to indicate the perceived health state from worst to best respectively.
Changes in the Modified Barthel Index (MBI) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  The MBI is an instrument used to assess the performance in Activities of Daily Living, and consists of 10 variables that reflect activities of daily living and mobility used to monitor functional status.
Changes in the Instrumental Activities of Daily Living Scale (IADL) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  The IADL Scale is used to assess more complex activities of daily living necessary for functioning in community living, such as handling finances and food preparation. It consists of 8 items which are summarily scored from zero (low functioning) to 8 (high functioning)
Changes in the Pittsburgh Sleep Quality Index (PSQI) scores at baseline, 3 months and 9 months | Baseline, 3 months, 9 months
  The PSQI is a self-report questionnaire that assesses sleep quality, and consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yee Tan, MMed(Psy), Principal Investigator — Associate Consultant
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared, in the interests of subject confidentiality

REFERENCES:
- [Background] Soga M, Gaston KJ, Yamaura Y. Gardening is beneficial for health: A meta-analysis. Prev Med Rep. 2016 Nov 14;5:92-99. doi: 10.1016/j.pmedr.2016.11.007. eCollection 2017 Mar. PMID 27981022
- [Background] Blake M, Mitchell G. Horticultural therapy in dementia care: a literature review. Nurs Stand. 2016 Jan 20;30(21):41-7. doi: 10.7748/ns.30.21.41.s44. PMID 26786461
- [Background] Noone S, Innes A, Kelly F, Mayers A. 'The nourishing soil of the soul': The role of horticultural therapy in promoting well-being in community-dwelling people with dementia. Dementia (London). 2017 Oct;16(7):897-910. doi: 10.1177/1471301215623889. Epub 2015 Dec 23. PMID 26701960
- [Background] Kamioka H, Tsutani K, Yamada M, Park H, Okuizumi H, Honda T, Okada S, Park SJ, Kitayuguchi J, Abe T, Handa S, Mutoh Y. Effectiveness of horticultural therapy: a systematic review of randomized controlled trials. Complement Ther Med. 2014 Oct;22(5):930-43. doi: 10.1016/j.ctim.2014.08.009. Epub 2014 Sep 1. PMID 25440385
- [Background] Annerstedt M, Wahrborg P. Nature-assisted therapy: systematic review of controlled and observational studies. Scand J Public Health. 2011 Jun;39(4):371-88. doi: 10.1177/1403494810396400. Epub 2011 Jan 27. PMID 21273226